CLINICAL TRIAL: NCT05291390
Title: A Phase 2a, Multi-centre, Randomised, Double-blinded, Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of Pyronaridine as an Add-on Therapy in Adults With Acute Lymphoblastic Leukemia and Acute Myeloid Leukemia
Brief Title: Pyronaridine in Acute Lymphoblastic Leukemia (ALL) and Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armaceutica, Inc. (Industry)
Collaborators: Uganda Cancer Institute (Other); African Center for Cancer Research and End of Life Care (ACREOL), Rwanda (Unknown); Ifakara Health Research and Development Centre (Other); Dalal Jamm Hospital, Dakar, Senegal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PND7351
Record Dates: First submitted 2021-10-07; First posted 2022-03-22 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-07

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphoblastic Leukemia (ALL)
Keywords: cancer; leukemia; phase 2; pyronaridine; oncology; treatment
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms; Leukemia | interventions — pyronaridine

STUDY DESIGN:
Intervention Model Description: The primary objective is the difference in survival lengths in days between the study arm receiving pyronaridine and the study arm receiving placebo as measured from the date of the first diagnosis of acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All capsules contain either pyronaridine or similar-appearing placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care treatment plus pyronaridine (Active Comparator): Standard of care treatment plus pyronaridine
  Interventions: Drug: Pyronaridine Tetraphosphate
- Standard of care treatment plus placebo (Placebo Comparator): Standard of care treatment plus placebo
  Interventions: Drug: Pyronaridine Tetraphosphate

INTERVENTIONS:
Drug: Pyronaridine Tetraphosphate — Via oral capsules.
  Other Names: Placebo

SUMMARY:
A Phase 2a clinical trial on up to n=200 male and female subjects 18 years and over who were diagnosed with acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL). Subjects are randomised in approximately a 1:1 ratio to receive standard of care treatment plus either pyronaridine (PND) or placebo. Quality of life parameters are measured. Visits include physical examinations, and blood draws for complete blood count with differential (CBC) and complete metabolic panel (CMP). Survival of subjects is tracked in Year 2.

DETAILED DESCRIPTION:
The primary objective is the difference in survival lengths in days between the study arm receiving pyronaridine and the study arm receiving placebo as measured from the date of the first diagnosis of acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL). Secondary objectives are differences between the active and placebo study arms in quality of life, laboratory data values and in the safety and tolerability of treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a diagnosis within 60 days of the time of study entry of either acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML). If the physician is a third-party physician, then the study site must obtain the subject's medical records from the clinic where the first diagnosis was made.
2. Subjects must be on standard of care therapy for ALL or AML. The standard of care therapy may be initiated at time of study entry.
3. Subjects must be 18 years of age or older, and male or female.
4. Subjects must weigh between 40kg and 90kg at time of study entry.
5. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) at least 14 days prior to study entry, for the duration of study participation, and at least 30 days after completion of drug administration. Women of child-bearing potential must agree to pregnancy tests for the duration of the study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the study subject should inform her investigator immediately.
6. Men must agree to always use a condom during intercourse for the duration of study participation, and for at least 30 days after completion of drug administration.
7. Subjects must have the ability to swallow size "0" gelatin capsules.
8. Subject must be willing to agree to and comply with all requirements of the study.
9. Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Subjects with malaria.
2. Subjects who are pregnant or nursing.
3. Subjects who have had major surgery within 30 days prior to study entry.
4. Subjects with active clinically significant infection or uncontrolled illness, except ALL or AML.
5. Subjects with evidence of chronic hepatitis B (HBV) infection.
6. Subjects with evidence or history of hepatitis C (HCV) infection.
7. Subjects with a prior or concurrent malignancy (basal cell carcinoma and squamous cell skin cancer are allowed).
8. Subjects with evidence of other disease or any concomitant medical or psychiatric problem which in the opinion of the investigator would put them at risk.
9. Subjects with a known hypersensitivity to pyronaridine tetraphosphate or compounds of similar chemical composition, or microcrystalline cellulose (MCC) the placebo agent.
10. Subjects who are receiving any other investigational agents or who have received any investigational medication within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in survival lengths to 1 year | 1 year
  The primary endpoint is the change in survival lengths in days between the study arm receiving pyronaridine and the study arm receiving placebo as measured from the date of the first known acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) diagnosis within 60 days of the time of study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Renato J Aguilera, PhD, Study Chair — Armaceutica, Inc.
Locations (1):
- Dalal Jamm Hospital, Guediawaye GOL SUD, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The Antimalarial Drug Pyronaridine Inhibits Topoisomerase II in Breast Cancer Cells and Hinders Tumor Progression In Vivo — https://pubmed.ncbi.nlm.nih.gov/30825052/
- See also: Pyronaridine exerts potent cytotoxicity on human breast and hematological cancer cells through induction of apoptosis — https://pubmed.ncbi.nlm.nih.gov/30395606/